CLINICAL TRIAL: NCT01534871
Title: The Effects of a 12-week Cardiovascular Rehabilitation Exercise Program on Inflammatory Markers and Traditional Coronary Artery Disease Risk Factors in Patients With Rheumatoid Arthritis
Brief Title: The Effects of Cardiac Rehabilitation on Cardiovascular Disease Risk in Rheumatoid Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDHA_NB_SG-2012
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Cardiac rehabilitation; Exercise; Systemic inflammation; Cardiovascular disease risk
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Subjects enrolled in the exercise arm will receive the study intervention.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Subjects in the control arm will receive standard of care (e.g. medication and medical supervision) for rheumatoid arthritis. These subjects will not participate in the exercise intervention.

INTERVENTIONS:
Behavioral: Exercise — Subjects will be enrolled in a 12-week community cardiac rehabilitation program. The program consists of two one hour exercise sessions per week and one one hour education session per week. For the exercise sessions the subjects will perform aerobic exercise at 60-80% of heart rate reserve. Education sessions will cover heart healthy eating, setting health-related goals, exercise, nutrition, healthy weight, medication, smoking cessation and stress/coping.
  Arms: Exercise

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease that affects approximately 1% of all Canadians. RA is associated with a higher rate of disease and death as well as a decreased life expectancy. Changes in death rates and life expectancy are mainly the result of an increased frequency of cardiovascular disease (CVD). The increase in CVD frequency is primarily attributable to accelerated atherosclerosis. It is believed that elevated levels of inflammation, which are characteristic of RA, play a key role in accelerated rate of CVD in RA patients. Thus, inflammation is considered a primary risk factor for CVD in RA patients. Interestingly, despite a better understanding of the relationship between RA and CVD and improved treatment for RA patients the death rate in RA population continues to increase. Thus, there is an immediate need to develop treatment strategies to reduce the risk of CVD associated with inflammation in the RA population.

Exercise is commonly used to reduce the risk of CVD. Preventative exercise programs are often offered as part of cardiac rehabilitation (CR) programs. These programs help patients modify CVD risk factors, improve physical capacity and decrease CVD risk. Studies also suggest that CR programs decrease levels of inflammation. Since RA patients have an elevated risk for CVD, which is primarily attributed to increased levels of inflammation, they are prime candidates for CR programs. However, RA patients are very rarely referred to CR programs. Thus, there is a lack of information regarding the effects of CR on RA patients. Thus studies are needed to determine whether CR modifies levels of inflammation and decreases CVD risk in RA patients. Therefore, the purpose of this study is to determine the effects of a 12-week standardized cardiac rehabilitation exercise program on systemic inflammation and CVD risk in individuals with RA. Specifically, this study will characterize the effects of a community based CR exercise program on systemic markers of inflammation (proinflammatory cytokines) and global CVD risk (Framingham risk profile) as well as the therapeutic effects of CR exercise on the severity of RA.

This study will help to clarify the mechanism(s) by which exercise impacts CVD risk in patients with inflammatory disease. In addition, the study will show how CR may benefit patients with inflammatory disease with respect to their ability to exercise, global risk for cardiovascular disease and quality of life.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease that impacts approximately 1% of all Canadians. RA is associated with increased mortality, decreased life expectancy and increased morbidity, which is primarily attributable to an increased risk of cardiovascular disease (CVD). Traditional risk factors (e.g. dyslipidemia, hypertension, physical inactivity, etc.) contribute, in part, to the elevated risk of CVD in individuals with RA. However, the higher incidence of CVD events in RA appears to be independent of the influence of traditional CVD risk factors. Non-traditional risk factors, such as inflammation, also contribute to the increased risk of CVD in RA patients. In fact, when traditional CVD risk factors and co-morbidities are controlled for in people with RA, markers of systemic inflammation confer a significant additional risk for CV death. This suggests that systemic inflammation significantly contributes to the increased risk of CVD in individuals with RA. Thus, there is an immediate need to develop intervention strategies to reduce the inflammatory mediated risk of CVD in the RA population.

One possible intervention that could be used to decrease CVD risk in RA patients is exercise. Exercise can modify both traditional (e.g. dyslipidemia) and non-traditional (e.g. inflammation) risk factors to decrease the risk of CVD. For patients with cardiac disease, clinical guidelines recommend regular exercise. For this, patients are referred to cardiac rehabilitation (CR) programs, where exercise represents the cornerstone of the program. The goal of these programs is modify CVD risk factors, improve physical capacity and decrease CVD risk. Thus, CR programs may offer a suitable therapeutic intervention to help decrease CVD risk in RA patients. However, RA patients are rarely referred to CR despite their increased risk of CVD. Thus, the effects of CR on inflammation and CVD risk in patients with RA remains unclear.

The purpose of this study is to examine the effects of a 12-week cardiac rehabilitation exercise program on systemic inflammation and CVD risk in individuals with RA. The specific objectives of the study are: 1) to determine whether it is feasible for RA patients to complete a 12-week high intensity CR exercise program, 2) examine the effects of a 12-week standardized CR exercise program on systemic markers of inflammation in individuals with RA, 3) to examine the effects of a 12-week standardized CR exercise program on CVD risk in individuals with RA and 4) to characterize the effects a 12-week standardized CR exercise program on the severity of the patient's RA and their functional ability.

This study is meant to be a pilot study that will help provide insight into the therapeutic effects of CR on inflammation and CVD risk in RA patients. Based on the results from this preliminary work, a larger scale study will be developed to evaluate the effects of exercise intensity on cardiovascular risk in patients with inflammatory disease as well as the effects of exercise on decision making for pharmacological intervention (e.g. statin therapy) in this population.

Methods:

Study Design: This pilot study is a randomized controlled study. Subjects will be randomly assigned to one of two groups: 1) control (CON) or 2) CR program with high intensity exercise (CRH). Outcome measures will be assessed at baseline (week-0) and post-intervention (week-13). The primary measures include CVD risk, levels of systemic inflammation and severity of RA. Secondary measures include weight, waist girth, resting heart rate, resting blood pressure (BP), lipid profile, fasting glucose, aerobic fitness, physical activity (PA) levels, functional ability, tobacco use and alcohol consumption.

Patient Screening: If the individual agrees to participate in the study, they will be asked if they use tobacco regularly and if they are a diabetic, have their BP measured and sent for routine blood work. Blood tests will be performed to determine the patient's lipid profile (total cholesterol, low density lipoprotein cholesterol, high density lipoprotein cholesterol and triglycerides). The patient's BP, answers to the aforementioned questions (e.g. tobacco, diabetes) and their lipid profile results will be used to calculate the patient's Framingham risk score, which estimates the 10-year CV risk of the patient.

Inclusion Criteria: Only those patients that 1) are 20 years of age or older 2) have RA fulfilling the American College of Rheumatology criteria, 3) have zero or more swollen joints, 4) are receiving stable pharmacotherapy (defined as greater than 3 months of unchanged antirheumatic drugs and greater than 1 month of unchanged nonsteroidal anti-inflammatory drugs), 5) have moderate risk of CVD as identified by the Framingham risk score, 6) are able to walk on treadmill or cycle on a stationary bike for 15 minutes and 7) are able to attend the Community Cardiovascular Hearts in Motion program (held in the Halifax Regional Municipality) will be asked to participate in the study. Any patients that meet the inclusion criteria, but are 1) known to have coronary, cerebral or peripheral artery disease, 2) taking statins, or 3) have one or more arthroplasties of weight bearing joints, will not be eligible to participate in the study.

Sample Size: The study will recruit 60 participants, 30 CON and 30 CRH..

Outcome measures: Variables pertaining to RA, CVD and PA will be measured in all subjects (CON, CRH) at two different time points during the study. Specifically, the subjects will be assessed at baseline (week-0) and then be reassessed post 12-week intervention (week-13). The post CR intervention assessment will be conducted 72 hours after the completion of the final exercise session. The variables that will be measured at week-0 and week-13 are listed in section B1e and the tools used to assess these outcomes are described below. Of note, the physicians/nurse conducting the assessments will be blinded in regards to which group the subject is assigned to.

RA Severity: Severity of RA will be determined using the American College of Rheumatology (ACR) response score. The ACR is a composite score based on 7 measures: 3 by an assessor (swollen joint, tender joint count and physician global status), 3 by the patient (function, pain and global status) and one acute phase measure (CRP). The ACR examination will be conducted by a rheumatologist (VB, Coinvestigator).

Aerobic Fitness: The subject's aerobic fitness will be determined based on the results from a stress test. All stress tests will be conducted by a cardiac research nurse. In brief, subjects will perform a graded exercise test (Bruce treadmill protocol) where speed and inclination of the treadmill increase every 3 minutes. The subject will be asked to exercise to volitional fatigue. Cardiac function will be monitored with a 12 lead ECG. The ECG data also will be used to determine if there is any evidence of cardiac disease (e.g. arrhythmia). Predictive equations developed for men and women will be used to calculate the subject's peak oxygen uptake. This value will represent the subject's aerobic fitness.

Physical Activity: The subject's current level of PA will be measured using the long form of the International Physical Activity Questionnaire. This questionnaire is suitable for use with clinical populations and has been used previously to quantify physical activity levels in RA patients.

Functional Ability: Functional status will be assessed using the short form of the Health Assessment questionnaire (HAQ). This is a self report questionnaire that is comprised of the HAQ disability index, HAQ patient global health status and the pain visual analog scale.

Blood Analysis: Blood samples will be drawn by either the research nurse or a physician. Samples will be processed at the local hospital to determine the subject's lipid profile, fasting glucose and CRP levels. Serum also will be extracted from the blood samples. Markers of systemic inflammation (cytokines) will be quantified in the serum samples. Specifically, tests will quantify levels of the proinflammatory cytokines IL-1α, IL-1β, IL-6, IL-17 and TNFα as well as the anti-inflammatory cytokines IL-4 and IL-10. Analysis will be performed at Dalhousie University (SG, PI) using a BioRad Bioplex Suspension Array System. All serum samples will be stored at -20°C until they are required for analysis.

Exercise Intervention:

Subjects will be randomly assigned to either the CON or CRH group. Subjects assigned to the CON will receive treatment for their RA that is considered standard care (e.g. pharmacotherapy), but will not be enrolled in the CR program. Subjects in the CON group will be asked to maintain their current level of PA during the course of the 12-week study. CON subjects will be given a log book to record their daily activity as well as report any significant changes in their PA level that occur during the study. Subjects assigned to the exercise group (CRH) will receive standard care for RA plus be enrolled in a CR program (Community Cardiovascular Hearts Motion Program, Halifax Regional Municipality, NS). The CR program is 12-weeks in duration and will be supervised by a nurse, a physiotherapist and a research assistant. The CR program is composed of one 60 minute education session per week and two 60 minute exercise sessions. The education sessions will be conducted by a multidisciplinary team of health professionals (nurse, physiotherapist and dietician). Topics covered include heart healthy eating, setting health-related goal, exercise, nutrition, healthy weight, smoking cessation and stress/coping. Some education sessions will be modified to better suit RA subjects (e.g. CVD medication session). The exercise sessions are based on standard of care for CVD patients. Exercise sessions will begin with a group a warm-up activity, followed by 45 minutes of aerobic activity and ending with a cool down. Aerobic activity will consist of walking/running on a treadmill, stepping exercise and/or cycling on a cycle ergometer. The subject will be encouraged to rotate through the various exercise machines (e.g. 15 minutes treadmill, 15 minutes cycle, 15 minutes stepper). All aerobic exercise will be performed at high intensity, which for the present study is defined as exercise that elicits a HR between 60-80% of heart rate reserve (HRR). Subjects will keep a log book for the duration of the program that details their exercise sessions. Subjects will record resting heart rate, type of exercise performed, duration of the exercise and HR during the exercise sessions. The subject also may add any relevant notes. All exercise sessions will be closely monitored by a nurse, physiotherapist and a research assistant. Prior to the initial CR exercise session target heart rates will be calculated for each subject based on the maximum HR achieved during their stress test. Subjects will be taught how to palpate radial and/or carotid pulse during the first week of the CR program. This will enable the subject to monitor and maintain their HR within the target HR zone while performing their aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Only those patients that 1) have RA fulfilling the American College of Rheumatology criteria, 2) have two or more swollen joints, 3) are receiving stable pharmacotherapy (defined as greater than 3 months of unchanged antirheumatic drugs and greater than 1 month of unchanged nonsteroidal anti-inflammatory drugs), 4) have moderate risk of CVD as identified by the Framingham risk score, 5) are able to walk on treadmill or cycle on a stationary bike for 15 minutes and 6) are able to attend the Community Cardiovascular Hearts in Motion program (held in the Halifax Regional Municipality).

Exclusion Criteria:

* Patients that are 1) diabetic, 2) have known coronary, cerebral or peripheral artery disease, 3) taking statins, or 4) have one or more arthroplasties of weight bearing joints will not be eligible to participate in the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Framingham risk score | Final measure week-13
  Equation used to predict global coronary heart disease risk. Factors used in the equation to predict risk include age, total cholesterol or LDL cholesterol, HDL cholesterol, blood pressure, history of diabetes and smoking history.
Levels of systemic inflammation | Final measure week-13
  Blood samples will be collected from the subjects and used to to quantify serum levels of proinflammatory cytokines (IL-1 alpha and beta, IL-6, IL-17 and TNF alpha) and anti-inflammatory cytokines (IL-4, IL-10).
Severity of rheumatoid arthritis | Final measure week-13
  Rheumatoid arthritis severity will be determined using the American College of Rheumatology (ACR) response score. The ACR is a composite score based on 7 measures: 3 by an assessor (swollen joint, tender joint count and physician global status), 3 by the patient (function, pain and global status) and blood work to measure rheumatoid factor (RF), anti-citrullinated protein antibodies (ACAP), c-reactive protein (CRP), and erythrocyte sedimentation rate (ESR)).

SECONDARY OUTCOMES:
Weight | Final measure week-13
Waist girth | Final measure week-13
  Waist girth will be measured at the level of the superior border of the iliac crest.
Resting heart rate | Final measure week-13
Resting blood pressure | Final measure week-13
Lipid profile | Final measure week-13
Aerobic fitness | Final measure week-13
  Aerobic fitness will be determined based a graded exercise test (Bruce treadmill protocol) where speed and inclination of the treadmill increase every 3 minutes. The subject will be asked to exercise to volitional fatigue. Cardiac function will be monitored with a 12 lead ECG to determine if there is any evidence of cardiac disease (e.g. arrhythmia). Predictive equations developed for men and women will be used to calculate the subject's peak oxygen uptake.
Physical activity level | Final measure week-13
  Physical activity will be measured using the long form of the International Physical Activity Questionnaire. This questionnaire is suitable for use with clinical populations and has been used previously to quantify physical activity levels in rheumatoid arthritis patients.
Functional ability | Final measure week-13
  Functional status will be assessed using the short form of the Health Assessment Questionnaire (HAQ). This is a self report questionnaire that is comprised of the HAQ disability index, HAQ patient global health status and the pain visual analog scale.
Smoking history | Final measure week-13
  Subjects will be asked whether they are currently a smoker or if they have smoked in the past 5 years.
Alcohol consumption | Final measure week-13
  Subjects will be asked to quantify there average weekly alcohol intake.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Giacomantonio, MD, Principal Investigator — Nova Scotia Health Authority; Scott A Grandy, PhD, Study Director — Dalhousie University
Locations (1):
- Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinze-Milne S, Bakowsky V, Giacomantonio N, Grandy SA. Effects of a 12-week cardiovascular rehabilitation programme on systemic inflammation and traditional coronary artery disease risk factors in patients with rheumatoid arthritis (CARDIA trial): a randomised controlled trial. BMJ Open. 2017 Dec 22;7(12):e018540. doi: 10.1136/bmjopen-2017-018540. PMID 29275344